CLINICAL TRIAL: NCT06017232
Title: The ParkinSANTÉlé Study: A Multicomponent Telerehabilitation Program to Improve Cardiovascular Health in People With Parkinson's Disease With a Clinical Diagnosis of Dysautonomia
Brief Title: Telerehabilitation for Dysautonomia in Parkinson's Disease
Acronym: PKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de Recherche sur le Vieillissement (CdRV) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20224665
Record Dates: First submitted 2023-08-08; First posted 2023-08-30 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: virtual rehabilitation; exercise; parkinsonism; cardiovascular; autonomic nervous system; cardiorespiratory; physical therapy; physiotherapy; physical activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: The study design is a pre-post without a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Group of participants receiving the hybrid telerehabilitation intervention
  Interventions: Other: Hybrid telerehabilitation program

INTERVENTIONS:
Other: Hybrid telerehabilitation program — The telerehabilitation program lasts 12 week (3 per week). The program includes aerobic, strength, coordination, balance, flexibility, and breathing exercises, in addition to educational components focused on disease management.
  This hybrid program incorporates both supervised and unsupervised sessions. A progressive approach from synchronous (supervised) to asynchronous (unsupervised) sessions is adopted.
  Each session is structured into 4 components: Warm-up; Muscle strengthening, coordination, and balance; Flexibility; and Breathing exercises.
  Participants are asked to maintain a log of their aerobic activity, recording details such as the type of activity, duration, and intensity. The aim is to align with the recommended aerobic physical activity guidelines (150 min/week). Weekly assessments are conducted to provide personalized guidance based on individual progress.
  Also, participants engage in weekly educational videos that cover a diverse range of PD-related topics.
  Other Names: OpenTera telerehabilitation

SUMMARY:
People diagnosed with Parkinson's Disease (PD) exhibit a combination of motor and non-motor symptoms, with the latter posing challenges in terms of identification and management. These non-motor symptoms tend to manifest before the motor symptoms and progressively worsen over time, significantly impacting the symptoms and everyday life activities of those affected. However, there remains a noticeable lack of scientific literature addressing the assessment and rehabilitation of cardiovascular dysautonomia in PD patients. Thus, our research aims to address this gap by pursuing the following objectives: 1) assess the feasibility, acceptability, and potential effectiveness of a hybrid telerehabilitation program designed to target cardiovascular health in individuals with Parkinson's disease; and 2) characterize cardiovascular dysautonomia using non-invasive measurements of cardiovascular and autonomic nervous system (ANS) function and self-reported symptom assessments.

DETAILED DESCRIPTION:
This pilot clinical trial employs mixed methods and aims to recruit 16 participants meeting the criteria of stage 1 to 3 Parkinson's disease according to the Hoehn and Yahr scale, aged 50 or above, under optimized drug therapy, having home internet access, and without exercise contraindications, but exhibiting cardiovascular dysautonomia based on positive clinical results from active orthostatic hypotension maneuver, with or without reported symptoms and/or SCOPA-AUT questionnaire score ≥ 2/3 items. The 12-week telerehabilitation program comprises three weekly sessions, encompassing different exercise modalities to improve walk capacity (aerobic, strength, balance, coordination, flexibility) and education on symptom management. A progressive increase in autonomy is implemented, starting with synchronous/asynchronous sessions of 3/0 in week 1 to 0/3 in week 12. Feasibility (recruitment, adherence, retention), acceptability (questionnaire, semi-structured interviews), and potential effectiveness on motor (walking, mobility, balance) and non-motor aspects (pain and cardiovascular dysautonomia) will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD (1 to 3 on Hoeh&Yahr)
* Patients under treatment with optimized drug therapy. Medication is stable for at least 1 month
* Patients with access to the internet
* Speaking French or English
* 50 years or older
* Patients having cardiovascular dysautonomia according to the clinical criteria: supine hypertension (SH) (≥140/90 mmHg) and/or orthostatic hypotension (OH) (a drop of systolic blood pressure ≥ 20 mmHg and/or diastolic blood pressure ≥ 10 mmHg during the active orthostatic hypotension test).

Exclusion Criteria:

* Major cognitive impairment (Montreal Cognitive Assessment, score ≤ 24)
* Neurological disorders other than PD
* Musculoskeletal or cardiopulmonary disorders preventing physical activity, contraindication to physical activity, or presence of a cardiac pacemaker.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the implementation | 12 weeks
  This will be evaluated by the percentage of participants that accepted to participate in the study (recruitment rate), percentage who completed the intervention (retention rate) and number of completed session in relation to the anticipated number of sessions (adherence).
Acceptability | 12 weeks
  The satisfaction of the participants will be evaluated with a questionnaire (14 questions). The questionnaire will assess patients' satisfaction with the professional, the services and the organization - Telemedicine Satisfaction. Qualitative open-ended questions will be used to determine appreciation and challenges encountered.
Dysautonomia Symptoms | 12 weeks
  Scale for Outcomes in Parkinson's disease for Autonomic symptoms (SCOPA-AUT) with maximum score 69, with the score for each item ranging from 0 (never experiencing the symptom) to 3 (often experiencing the symptom).
Impact of dysautonomia symptoms | 12 weeks
  Orthostatic Hypotension Questionnaire (OHQ): The questionnaire is divided into 2 parts: Part I, Symptom Assessment (OHSA), consisted of 6 questions, each rat-ing the intensity of one characteristic symptom [ 1. Dizziness, lightheadedness, feeling faint, or feeling Iike you might black out; 2. Problems with vision (blurring, seeing spots, tunnel vision, etc.); 3. Generalized weakness; 4. Fatigue; 5. Trouble concentrating; 6. Head/neck dis-comfort] and Part Il, Daily Activity Scale (OHDAS), consisted of 4 questions that assessed the impact of NOH symptoms on daily activities.
  Items scored on an 11-point scale (0 to 10), with O indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference. The composite OHQ score is calculated by averaging the OHSAS and the OHDAS.
Exercise capacity | 12 weeks
  Six-minute walk test (performance and physiological responses)

SECONDARY OUTCOMES:
Severity of pain and impact on functioning | 12 weeks
  Brief Pain Inventory: Participants are asked to rate their current symptoms, their average experiences of pain, and the minimum and maximum intensities of their symptoms on scales that range from 0 to 10. A total pain severity score can be found by averaging these items or a single item can be treated as the primary outcome measure.
Type of pain | 12 weeks
  Neuropathic pain DN4 Questionnaire: Items are scored based on a yes (1 point) /no (0 points) answer. This leads to a score range of 0-10 when the symptoms (range 0-7 points) as well as the signs (range 0-3 points) items are included.
Perceived quality of life | 12 weeks
  Parkinson's Disease Questionnaire 8 items (PDQ-8, scored 0-32, higher score indicating the worst quality of life)
Lower-limb function | 12 weeks
  Lower Extremity Functional Scale (LEFS, scored 0-32, higher score indicating less difficulty)
Mobility in the community | 12 weeks
  Life-space mobility (French-Canadian version) (partial scores are summed to produce a composite score 0-120, higher score indicating more mobility)
Mobility | 12 weeks
  Timed Up and Go
Balance | 12 weeks
  Berg balance scale (scored 0-56, higher score indicating more balance)
Walking capacity | 12 weeks
  10-meter walk test
Lower-limb strength and power | 12 weeks
  5-repetition sit to stand test
Cardiovascular health | 12 weeks
  24-hour ambulatory blood pressure monitoring (Mobil-O-Graph® 24hr ABPM) (systolic and diastolic blood pressure)
Sympathetic nervous innervation of the skin | 12 weeks
  Electrodermal activity (Galvanic skin response) with PowerLab ADInstruments: Results are presented as the difference between the maximum of the electrodermal response (or of sweating, therefore of skin conductivity) and the minimum of the electrodermal response (delta values).
Autonomic modulation | 12 weeks
  Heart rate variability (HRV) (supine 6 minutes and upright position 6 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Livia Pinheiro Carvalho, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada